CLINICAL TRIAL: NCT02588079
Title: Internet-Based Cognitive Behavioral Therapy for Children With Dental Anxiety- A Randomized Controlled Trial
Brief Title: Internet-Based Cognitive Behavioral Therapy for Children With Dental Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Shervin Shahnavaz, Psychologist, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KIPED20151008
Record Dates: First submitted 2015-10-22; First posted 2015-10-27 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Dental Anxiety
Keywords: Dental Fear; Dental Phobia; Internet based cognitive behavioral therapy; specific phobia; children and adolescents anxiety; Self Efficacy
MeSH Terms: conditions — Phobia, Specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based cognitive behavioral therapy (Experimental): The treatment program consists of 12 modules that are offered during 12 weeks on Internet. Modules consist of parental education, psycho-education for the children, exposure, cognitive restructuring and home exercises. A psychologist guides parents and children through the treatment with continuous contact using the message function on the Internet platform that is used.
  Interventions: Behavioral: Internet-based cognitive behavioral therapy
- Wait list (No Intervention): Participants are not offered any active controlled psychological interventions but have free access to dental health services, which could involve exposure and other behavioral strategies applied by dental staff.

INTERVENTIONS:
Behavioral: Internet-based cognitive behavioral therapy
  Arms: Internet-based cognitive behavioral therapy

SUMMARY:
The purpose of this study is to determine whether internet-based cognitive behavioral therapy (ICBT) is effective in the treatment of children and adolescents with dental anxiety. The investigators hypothesis is that children and adolescents who have been offered ICBT show significant better performance on outcome measures compared with patients in control group.

ELIGIBILITY:
Inclusion Criteria:

* The participant is between 8-15 years of age
* The patient and parents agree to participate in the research project
* A diagnosis of specific phobia (dental anxiety or intraoral needle phobia) can be established by a psychologist according to the Diagnostic and Statistical Manual of Mental Disorders, 4th. Edition. The internet parent version of Development and Well-Being Assessment (Dawba) and Kiddie Sads (phobic disorders supplement) are used.
* The patient and parents have sufficient language skills in Swedish to manage the treatment and questionnaires
* Have regularly access to computer and the internet
* Have the time, the possibility and motivation to work and practice with ICBT 3 hours each week in 12 weeks
* Parents agree to at least book three visits at the dentist during the 12 weeks treatment
* Parents agree to exposure for intraoral injection at the dentist even if the child does not need dental treatment but suffers from injection phobia

Exclusion Criteria:

* Full points on both child and parent versions of the picture guided behavioral approach test. A maximum score of 17 means that both the child and the parent assess that the child can manage the most challenging situations in dentistry
* A score of 31 or less on both children and parent version of CFSS-DS and do not fulfill criteria for intra-oral injection phobia
* Already have or according to DAWBA and/or telephone interview by psychologist likely to fulfill criteria for a neurodevelopmental disorder diagnosis
* Other psychiatric disorders such as severe depression, eating disorder or self harm behavior that need treatment prior to dentistry related specific phobia
* The participant is undergoing or has planned psychiatric/ psychological examination
* The participant has current/planed psychological treatments
* Stressful life experiences during the past 12 months, such as divorce in the family, somatic illness that parent or the psychologist see as an obstacle in the treatment
* Have received cognitive behavioral treatment for dental anxiety or needle phobia during the past three years

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Picture guided behavioral approach test, child version | post treatment(12 weeks), and follow up (12 months after posttreatment)
  Measures changes in self-estimated ability to manage 17 dental situations, showing realistic images from dental care.
Picture guided behavioral approach test, parent version | post treatment(12 weeks), and follow up (12 months after posttreatment)
  Measures changes in the child´s ability to manage dental situations according to a parent. The test shows 17 realistic images from the dental care.

SECONDARY OUTCOMES:
Self-Efficacy Questionnaire for Phobic Situations ( dentistry adapted version ) | post treatment(12 weeks), and follow up (12 months after posttreatment)
  Measure changes in child's dentistry related self efficacy
Children's Fear Survey Schedule - Dental Subscale (child version) | post treatment(12 weeks), and follow up (12 months after posttreatment)
  Measures changes in the child's dental anxiety
Children's Fear Survey Schedule - Dental Subscale (parent version) | post treatment(12 weeks), and follow up (12 months after posttreatment)
  Measures changes in the child's dental anxiety according to one of the parents
Kiddie Sads (phobic disorders supplement) | post treatment(12 weeks), and follow up (12 months after posttreatment)
  The phobic disorders supplement of Kiddie Sads diagnostic interview (Version 1.0 of October 1996) is performed by a psychologist through a telephone interview. The outcome is used to investigate whether the participant fulfill the diagnostic criteria for dentistry related specific phobia according to DSM 4.

OTHER OUTCOMES:
Parental Self-Efficacy Questionnaire for Dental Anxiety | post treatment(12 weeks), and follow up (12 months after posttreatment)
  Measure changes in dentistry related parental self efficacy
Children's Negative Cognitions in Dentistry | post treatment(12 weeks), and follow up (12 months after posttreatment)
  Measure changes in children's dentistry related negative thoughts.
Injection Phobia Scale for Children | post treatment(12 weeks), and follow up (12 months after posttreatment)
  Measure changes in children's degree of anxiety related to injection

CONTACTS AND LOCATIONS:
Overall Officials: Shervin Shahnavaz, PhD, Principal Investigator — Department of Dental Medicine, Karolinska Institutet
Locations (1):
- Department of Dental Medicine, Stockholm, Huddinge, Sweden

REFERENCES:
- [Background] Shahnavaz S, Hedman-Lagerlof E, Hasselblad T, Reuterskiold L, Kaldo V, Dahllof G. Internet-Based Cognitive Behavioral Therapy for Children and Adolescents With Dental Anxiety: Open Trial. J Med Internet Res. 2018 Jan 22;20(1):e12. doi: 10.2196/jmir.7803. PMID 29358158
- [Background] Shahnavaz S, Hedman E, Grindefjord M, Reuterskiold L, Dahllof G. Cognitive Behavioral Therapy for Children with Dental Anxiety: A Randomized Controlled Trial. JDR Clin Trans Res. 2016 Oct;1(3):234-243. doi: 10.1177/2380084416661473. Epub 2016 Aug 15. PMID 29417092
- [Background] Shahnavaz S, Rutley S, Larsson K, Dahllof G. Children and parents' experiences of cognitive behavioral therapy for dental anxiety--a qualitative study. Int J Paediatr Dent. 2015 Sep;25(5):317-26. doi: 10.1111/ipd.12181. Epub 2015 Jul 4. PMID 26147012
- [Derived] Schibbye R, Hedman-Lagerlof E, Kaldo V, Dahllof G, Shahnavaz S. Internet-Based Cognitive Behavioral Therapy for Children and Adolescents With Dental or Injection Phobia: 1-year Follow-Up Assessment. JMIR Pediatr Parent. 2025 Sep 17;8:e80376. doi: 10.2196/80376. PMID 40962319
- [Derived] Schibbye R, Hedman-Lagerlof E, Kaldo V, Dahllof G, Shahnavaz S. Internet-Based Cognitive Behavioral Therapy for Children and Adolescents With Dental or Injection Phobia: Randomized Controlled Trial. J Med Internet Res. 2024 Feb 21;26:e42322. doi: 10.2196/42322. PMID 38381476
- See also: Registration website — http://ki.se/dentmed/kbt